CLINICAL TRIAL: NCT04073680
Title: A Phase 1b/2 Study of Serabelisib in Combination With Canagliflozin in Patients With Advanced Solid Tumors With PIK3CA or KRAS Mutations
Brief Title: A Phase 1b/2 Study of Serabelisib in Combination With Canagliflozin in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Petra Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT06-01
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Endometrial Cancer; Lung Cancer; Colo-rectal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Lung Neoplasms; Colonic Neoplasms; Head and Neck Neoplasms | interventions — serabelisib; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Serabelisib (Experimental): Part 1 is dose escalation of Serabelisib Cohort 1 = 600mg; Cohort 2 = 900mg; Cohort 3 = 1200mg
  Part 2 is expansion of mutational cohorts with selected dose as follows:
  Cohort 4 = PIK3CA-mutated breast cancer; Cohort 5 = PIK3CA-mutated Non breast cancer; Cohort 6 = KRAS mutated
  Interventions: Drug: Serabelisib; Drug: Canagliflozin 300mg

INTERVENTIONS:
Drug: Serabelisib — Subjects will be dosed with Serabelisib on 3 consecutive days a week in a 28 day cycle until tumor progression. in combination with Canagliflozin 300mg, both are oral medications
Drug: Canagliflozin 300mg — All subjects will be dosed with 300 mg canagliflozin in combination with serabelisib
  Other Names: Invokana

SUMMARY:
This study aims to test the hypothesis that combining serabelisib, a PI3K alpha isoform inhibitor, with an SGLT2 inhibitor, canagliflozin will improve efficacy in the treatment of patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study aims to test the hypothesis that controlling the glucose/insulin feedback will enhance the efficacy of PI3K inhibition in treating solid tumors. The treatment consists of serabelisib, a PI3K alpha isoform (PI3Kα) inhibitor, combined with the sodium-glucose cotransporter-2 (SGLT2) inhibitor canagliflozin. The study will assess the safety and efficacy of the combination in adult patients with advanced solid tumors harboring mutations that may be dependent on PI3Kα activity: PIK3CA mutations and KRAS mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed locally advanced or metastatic solid tumors.
2. Have a tumor harboring a mutation in PIK3CA or KRAS genes.
3. Have received prior therapy and have recurrent or persistent disease without standard therapies available, or are ineligible to receive standard therapies.
4. Have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
5. Have Eastern Cooperative Oncology Group performance status (ECOG PS) of ≤2
6. Have adequate organ function.
7. Have adequate birth control during the course of the study.

12. Are able to receive canagliflozin

Exclusion Criteria:

1. Diagnosis of primary brain tumor
2. Untreated brain metastasis or history of leptomeningeal disease
3. Have received prior chemotherapy within 28 days or other anticancer agents within 28 days of 5 half lives (whichever is the shorter duration) before the first administration of study drug. The exception is patients in Cohort 4 (PIK3CA-mutated breast cancer) are allowed to receive ongoing endocrine therapy.
4. Have diabetes mellitus requiring insulin therapy
5. Have diabetes mellitus requiring insulin secretagogue therapy
6. Have poorly controlled diabetes mellitus defined as glycosylated hemoglobin A1c (HbA1c) >7.5%
7. Have a secondary malignancy requiring therapy or are unstable without therapy.
8. Known impaired cardiac function or clinically significant cardiac disease.
9. Myocardial infarction or unstable angina within 6 months before the first administration of study drug.
10. Pregnant (positive serum pregnancy test) or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse Events | 30 days after last dose
  Safety of serabelisib in combination with canagliflozin as evaluated by incidence of drug-related adverse events (AEs), serious adverse events (SAEs), adverse events leading to discontinuation, deaths and clinical laboratory test abnormalities.
Rate of Laboratory Abnormalities | 30 days after last dose
  Safety of serabelisib in combination with canagliflozin as evaluated by incidence of clinical laboratory abnormalities
Dose confirmation | 6 months
  To confirm the appropriate dose of serabelisib to be coadministered with canagliflozin
Tumor Assessments by RESIST | 2 years
  To assess efficacy of serabelisib in combination with canagliflozin in patients with solid tumors with PIK3CA or KRAS mutations

SECONDARY OUTCOMES:
Cmax Pharmacokinetic assessment | Day 1 and 8 of Cycle 1: pre-dose and then post-dose at 1.5 hours, 3 hours, 6 hours, 9 hours, 12 hours, and 24 hours
  Maximum observed plasma concentration (Cmax) of serabelisib
Tmax Pharmacokinetic assessment | Day 1 and 8 of Cycle 1: pre-dose and then post-dose at 1.5 hours, 3 hours, 6 hours, 9 hours, 12 hours, and 24 hours
  Time of maximum observed plasma concentration (Tmax) of serabelisib
AUC Pharmacokinetic assessment | Day 1 and 8 of Cycle 1: pre-dose and then post-dose at 1.5 hours, 3 hours, 6 hours, 9 hours, 12 hours, and 24 hours
  Area under the plasma concentration time curve in the dosing interval AUC of serabelisib

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yu, MD, Study Director — Petra Pharma

IPD SHARING:
Plan to Share IPD: No